| Project Title: Use | r Evaluation o | of the Gui | ide To Go | als Applica | tion - a | Care C | Coordination | Tool to | Translate |
|---|---|---|---|---|---|---|---|---|---|
| | ADA Clinical | Standard | ls of Care | for Childre | en With | T2D Ir | nto Practice | | |

NCT Number: NCT03926598

Date: December 13, 2022

## **Statistical Analysis Plan**

Percentages of completion of the usability tasks were calculated for each group and as a whole. In total, five groups were analyzed (1. Patients/caretakers 2. Front-desk staff 3. Nurses 4. Certified Diabetes Educators) and the following tasks listed below were analyzed for each group. Additionally, qualitative analyses were used to analyze the results from the interviews and questionnaires.

# Tasks to be completed by group:

- 1. Patient and/or Family Member
  - a. On the Patient Login Screen, log in using your last name and session ID provided by the research team on the Surveys Screen.
  - b. Click on a pending survey when the survey opens.
  - c. Respond to the survey submit the survey log out of the Guide-Goals Application

#### 2. Front Desk Staff

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patient Screen.
- b. Add a new patient on the Edit Patient Screen.
- c. Add the Diabetes Family Responsibility Questionnaire on the Edit Patient Screen.
- d. Create a survey access code to share with the patient

#### 3. Nurse

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen.
- b. Choose patient Will Owens on the Visit Status screen.
- c. Change HbA1C value to 10% on the Visit Status screen.
- d. Change Nephropathy evaluation to Abnormal log out of Guide to Goals application.

### 4. Certified Diabetes Educator

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen.
- b. Choose patient Will Owens on the Visit Status Screen.
- c. Add comments needs to be followed up regarding ketosis education in the comments for provider text box on the Visit Status Screen.
- d. Add a goal for the patient log out of Goals-to-Guide application.